CLINICAL TRIAL: NCT02815462
Title: Impact of Implementing a Real Time Frequent Admitter Risk Score (FAM-FACE-SG) on Readmission Rates: a Pragmatic Cluster Randomised Controlled Trial (RCT).
Brief Title: Impact of Implementing a Real Time Frequent Admitter Risk Score (FAM-FACE-SG) on Readmission Rates
Acronym: FAMFACESGRCT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to secure grant funding
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SGH_OIC_FAMFACESG/5/2016
Record Dates: First submitted 2016-06-20; First posted 2016-06-28 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Patient Readmission
Keywords: Frequent hospital admissions; Risk stratification; Readmissions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): FAM-FACE-SG risk score + decision making algorithm
  Interventions: Other: FAMFACESG
- Control (Active Comparator): Usual Care
  Interventions: Other: Control

INTERVENTIONS:
Other: FAMFACESG — - PNs will receive the FAM-FACE-SG FA risk scores for frequent admitters admitted to their ward.
  Arms: Intervention
Other: Control — - Usual hospital Care
  Arms: Control
Other: FAMFACESG — - PNs will be instructed to prioritize intervention of frequent admitters for intervention based on the FA risk score.
  Arms: Intervention
Other: FAMFACESG — * For high and moderate risk patients who do not require transitional home care (THC), PN will do the case management and follow up.
  * For high and moderate risk patients & have complex nursing and / or high functional needs, PNs will refer these patients for THC.
  * For mild risk patients, PNs will refer them to care coordinator.
  Arms: Intervention
Other: FAMFACESG — - For low risk patients, PNs will continue usual hospital care.
  Arms: Intervention

SUMMARY:
In an earlier study using electronic health records (EHR), the investigators have identified nine factors to be significantly associated with FA risk. These nine predictors include Furosemide intravenous 40 milligrams or more; Admissions in the past one year; Medifund status; Frequent emergency department use; Anti-depressants treatment in past one year; Charlson comorbidity index; End Stage Renal Failure on dialysis; Subsidized ward stay and Geriatric patient. The investigators have combined these nine predictors into the FAM-FACE-SG score for FA risk (defined as 3 or more inpatient admissions in the following 12 months). The FAM-FACE-SG risk score has the advantage of being deployed in our hospital's enterprise data repository known as Electronic Health Intelligence System or eHINTs for short, on a real-time or near real-time basis. On a daily basis, data from multiple data sources are extracted, transformed and loaded onto the eHINTS system. The system can be programmed to run every midnight to provide risk scores the following morning for patients admitted the previous day.

In this trial, the intervention is to combine the FAM-FACE-SG risk score in addition to a decision making algorithm to guide referrals to various transitional care services based on needs assessment on nursing and function. The primary objective is to evaluate the impact of our intervention in improving healthcare utilization (hospital readmissions, emergency department (ED) attendances, length of stay up to 90 days post-discharge).

DETAILED DESCRIPTION:
In an earlier study using electronic health records (EHR), The investigators have identified nine factors to be significantly associated with FA risk. These nine predictors include Furosemide intravenous 40 milligrams or more; Admissions in the past one year; Medifund status; Frequent emergency department use; Anti-depressants treatment in past one year; Charlson comorbidity index; End Stage Renal Failure on dialysis; Subsidized ward stay and Geriatric patient. The investigators have combined these nine predictors into the FAM-FACE-SG score for FA risk (defined as 3 or more inpatient admissions in the following 12 months). The FAM-FACE-SG risk score has the advantage of being deployed in our hospital's enterprise data repository known as Electronic Health Intelligence System or eHINTs for short, on a real-time or near real-time basis. On a daily basis, data from multiple data sources are extracted, transformed and loaded onto the eHINTS system. The system can be programmed to run every midnight to provide risk scores the following morning for patients admitted the previous day.

In this trial, the intervention is to combine the FAM-FACE-SG risk score in addition to a decision making algorithm to guide referrals to various transitional care services based on needs assessment on nursing and function. The primary objective is to evaluate the impact of our intervention in improving healthcare utilization (hospital readmissions, emergency department (ED) attendances, length of stay up to 90 days post-discharge).

The aims of this cluster RCT are to: (1) evaluate the impact of implementing the FAM-FACE-SG risk score in addition to a decision making algorithm to guide Patient Navigator (PN) referrals to various transitional care services based on needs assessment on nursing and function on improving healthcare utilization (hospital readmissions, emergency department (ED) attendances, length of stay up to 90 days post-discharge); (2) measure the implementation of the risk score (Fidelity of the PNs in adhering to the protocol in recruiting patients according the score priority; Referral rate of the PNs to various transitional care services; Qualitative feedback from PNs on the perceived benefits and behavior change after receiving the scores); (3) conduct an economic analysis of the cost-benefit of implementing the risk score.

ELIGIBILITY:
Inclusion Criteria:

* Singapore General Hospital wards with patient navigators
* Patients who are frequent admitters (defined as 3 or more hospital admissions in the preceding 12 months)

Exclusion Criteria:

* Haematology, Oncology, Emergency department, obstetrics and neonatology wards

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
90-day readmission rate | 90 days

SECONDARY OUTCOMES:
30-day readmission rate | 30 days
30-day ED attendance rate | 30 days
90-day ED attendance rate | 90 days
index hospital admission length of stay | 90 days
cumulative length of stay 90 days after index hospital discharge | 90 days
Fidelity of the PNs in following the protocol in recruiting patients according the score priority | 90 days
Proportion of high and medium risk patients recruited in both intervention and control groups | 90 days
Referral rate of the PNs to various transitional care services | 90 days
Qualitative feedback from PNs on the perceived benefits and behaviour change after receiving the scores | 1 year
  Questionnaire survey

CONTACTS AND LOCATIONS:
Overall Officials: Lian Leng Low, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kripalani S, Theobald CN, Anctil B, Vasilevskis EE. Reducing hospital readmission rates: current strategies and future directions. Annu Rev Med. 2014;65:471-85. doi: 10.1146/annurev-med-022613-090415. Epub 2013 Oct 21. PMID 24160939
- [Result] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721
- [Result] Robst J. Developing Models to Predict Persistent High-Cost Cases in Florida Medicaid. Popul Health Manag. 2015 Dec;18(6):467-76. doi: 10.1089/pop.2014.0174. Epub 2015 Jun 23. PMID 26102363
- [Result] Longman JM, I Rolfe M, Passey MD, Heathcote KE, Ewald DP, Dunn T, Barclay LM, Morgan GG. Frequent hospital admission of older people with chronic disease: a cross-sectional survey with telephone follow-up and data linkage. BMC Health Serv Res. 2012 Oct 30;12:373. doi: 10.1186/1472-6963-12-373. PMID 23110342
- [Result] Low LL, Vasanwala FF, Ng LB, Chen C, Lee KH, Tan SY. Effectiveness of a transitional home care program in reducing acute hospital utilization: a quasi-experimental study. BMC Health Serv Res. 2015 Mar 14;15:100. doi: 10.1186/s12913-015-0750-2. PMID 25888830